CLINICAL TRIAL: NCT03992287
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Hydrolysed Red Ginseng Extract on Dry Eye
Brief Title: Efficacy and Safety of Hydrolysed Red Ginseng Extract on Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, You, In Cheon, Professor of ophthalmology, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GH-DE-HR
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolysed Red Ginseng Extract (Experimental): 10 ml/day, 2.4g/day for 12 weeks
  Interventions: Dietary Supplement: Hydrolysed Red Ginseng Extract
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolysed Red Ginseng Extract — 10 ml/day, 2.4g/day for 12 weeks
  Arms: Hydrolysed Red Ginseng Extract
Dietary Supplement: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Hydrolysed Red Ginseng Extract extract on dry eye.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. 46 subjects were randomly divided into Hydrolysed Red Ginseng extract 10ml or placebo group. The investigators measured Ocular Surface Disease Index, tear break-up time, Visual analog scale, Schirmer's test, meibomian gland test and Fluorescein staining.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 19years
* Ocular Surface Disease Index score is 13 scores and more at a screening
* Tear Break-Up Time is 10 seconds less or those who have positive in ocular staining test at a screening
* After fully hearing and fully understanding this clinical trials, those who agree to voluntarily decide to participate and to comply with the notice

Exclusion Criteria:

* Those who have a body mass index(BMI) of less than 18.5 kg / m^2 or greater than 35 kg / m^2 at the screening
* Those who have clinically significant acute or chronic ophthalmologic, cardiovascular system, endocrine, immune, respiratory, liver biliary system, renal and urinary tract, neuropsychiatry, musculoskeletal, inflammatory and hematologic and gastrointestinal disorders
* Those who couldn't control diabetes at screening
* Those with acute eye infections or inflammation within 1 month before screening
* Those who have ophthalmic surgery within 3 months before screening
* Those who use contact lens 1 month before screening
* Those who take a medication or health function food that affects your promotion of dry eye within 1 month prior to the screening
* Those who have received antipsychotic medication within 3 months before screening
* Those who alcoholic or drug abuse suspected
* Those who participated in other clinical trials within 3 months before screening
* Laboratory test by showing the following results

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breastfeeding
* Those who don't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in the study because of Laboratory test results, etc.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Ocular Surface Disease Index | 12 weeks
  A questionnaire which is Ocular Surface Disease Index consisted of 12 questions each of which included visual symptoms, visual work status, and environmental factors.
  The Ocular Surface Disease Index scores are ranged from 0 to 100, and the high score is the more severe the symptoms. The Ocular Surface Disease Index score is calculated as follows.
  : (Sum of all items answered × 25) / total number of questions answered
Changes of tear break-up time | 12 weeks
  The tear break-up time test measures the time in seconds. The time is from the last blinking to the point of tear layer defect or streak-like defect after blinking the eye with 1% of fluorescein.
  10 seconds or more as normal, between 5 and 10 seconds as mild dry eye syndrome, and 5 seconds or less as severe dry eye syndrome.

SECONDARY OUTCOMES:
Changes of Visual analog scale | 12 weeks
  The Visual Analog Scale(VAS) score is 0 point for no symptom, 10 points for the most severe symptom, and the patient is asked to mark the degree of subjective pain symptoms as an integer.
Changes of Schirmer's test | 12 weeks
  Schirmer's test determines whether the eye produces enough tears to keep it moist. This test is used when a person experiences very dry eyes or excessive watering of the eyes. It poses no risk to the subject. A negative (more than 10 mm of moisture on the filter paper in 5 minutes) test result is normal. Both eyes normally secrete the same amount of tears.
Changes of meibomian gland test | 12 weeks
  Meibomian gland test evaluate 8 Meibum of the upper middle eyelid or lower middle eyelid. The Meibum quality score and the Meibum expressibility score are evaluated as follows.
  * Meibum quality score 0 = clear fluid
    1. = cloudy fluid
    2. = cloudy particulate fluid(with debris)
    3. = inspissated (opaque),like toothpaste
  * Meibum expressibility score 0 = all glands expressible
    1. = three to four glands expressible
    2. = one to two glands expressible
    3. = no glands expressible
Changes of Fluorescein staining | 12 weeks
  Fluorescein staining was evaluated by staining with 1% fluorescein (1% sodium fluorescein 1 μL volume), and then assessed for damage after corneal and conjunctival staining. The degree of staining of the cornea is divided into 5 sections according to the NEI scale, and each section is judged as 0 ~ 3 scores. It is judgement the degree of severity from 0 to 15 scores per eye. The degree of conjunctival staining is divided into six sections per eye, and each section is scored 0 to 3 scores total 0 ~ 18 scores.

CONTACTS AND LOCATIONS:
Overall Officials: In Cheon You, M.D., Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea